CLINICAL TRIAL: NCT00882518
Title: A 6-Week, Multi-centre, Double-blind, Double-dummy, Chlorpromazine-Controlled Randomised Study to Evaluate the Efficacy and Safety of Quetiapine Fumarate Extended-Release in the Treatment of Schizophrenic Patients With Acute Episode
Brief Title: Efficacy and Safety of Quetiapine Fumarate in the Treatment of Schizophrenic Patients
Acronym: ESPRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1444C00008
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: Quetiapine Fumarate (SEROQUEL) Extended-Release (XR); qualified PANSS assessment
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Chlorpromazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) (Experimental): Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) extended-release (300 mg/1st day, 600 mg/2nd day, 400 or 600 or 800 mg/3-42 day)
  Interventions: Drug: Quetiapine Fumarate (SEROQUEL) Extended-Release (XR)
- 2-Chlorpromazine (Active Comparator): Chlorpromazine (50 or 100 mg/1st day; 100-200 mg/2nd day; 150-300 mg/3rd day; 200-400 mg/4th day; 300 or 400 or 500 or 600 mg/5-42 days)
  Interventions: Drug: Chlorpromazine

INTERVENTIONS:
Drug: Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) — 200 mg or 300 mg, oral, single dose
  Other Names: Seroquel_XR (Quetiapine Fumarate XR)
  Arms: 1-Quetiapine Fumarate (SEROQUEL) Extended-Release (XR)
Drug: Chlorpromazine — 50 mg, oral, double dose
  Arms: 2-Chlorpromazine

SUMMARY:
The primary objective of this study is to evaluate the efficacy of quetiapine fumarate extended-release (XR) used as mono-therapy, administered once daily, in the treatment of schizophrenic patient with acute episode.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia diagnosis
* Provision of written informed consent before initiation of any study

Exclusion Criteria:

* AIDS and hepatitis B
* History of seizure disorder
* Hospitalisation for schizophrenic more than 1 month immediately before enter into study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niufan Gu, Principal Investigator — Shanghai Mental Health Center; Michael Castiglione, Study Director — AstraZeneca
Locations (11):
- China (11):
  - Research Site, Hunan, Changsha
  - Research Site, Guangzhou, Guangdong
  - Research Site, Baoding, Hebei
  - Research Site, Harbin, Heilongjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Xi’an, Shanxi
  - Research Site, Kunming, Yunnan
  - Research Site, Beijing
  - Research Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 388 patients from 11 sites were randomised into Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) group or chlorpromazine group.
Groups:
- Quetiapine Fumarate (SEROQUEL) Extended-Release (XR): Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) was administered orally, once daily in the evening. The initial dose was 300 mg. This dose was adjusted on Day 2 to 600 mg, from Day 3 to Day 42, the dose of Quetiapine fumarate XR could be adjusted at 400 mg/day, 600 mg/day, or 800 mg/day at the investigator's discretion.
- Chlorpromazine: Chlorpromazine was administered orally, twice daily. The initial dose was 50 mg to 100 mg. This dose was adjusted on Day 2 from 100 to 200 mg, on Day 3 from 150 to 300 mg, and Day 4 from 200 to 400 mg. From Day 5, the dose of chlorpromazine could be adjusted at 300 mg/day, 400 mg/day, 500 mg/day, or 600 mg/day at the investigator's discretion.
Period: Overall Study
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Started | 196 | 192
Completed | 158 | 148
Not Completed | 38 | 44
Not completed — Adverse Event | 9 | 18
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Lack of Efficacy | 12 | 9
Not completed — Severe non-compliance to protocol | 3 | 1
Not completed — Incorrect enrolment | 4 | 2
Not completed — Central lab closure for National day | 1 | 0
Not completed — Allocating random number by mistake | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Seroquel_XR: Quetiapine fumarate XR was administered orally, once daily in the evening. The initial dose was 300 mg. This dose was adjusted on Day 2 to 600 mg, from Day 3 to Day 42, the dose of Quetiapine fumarate XR could be adjusted at 400 mg/day, 600 mg/day, or 800 mg/day at the investigator's discretion. Full analysis set (FAS) population used for baseline characteristics
- Chlorpromazine: Chlorpromazine was administered orally, twice daily. The initial dose was 50 mg to 100 mg. This dose was adjusted on Day 2 from 100 to 200 mg, on Day 3 from 150 to 300 mg, and Day 4 from 200 to 400 mg. From Day 5, the dose of chlorpromazine could be adjusted at 300 mg/day, 400 mg/day, 500 mg/day, or 600 mg/day at the investigator's discretion. Full analysis set (FAS) population used for baseline characteristics
- Total: Total of all reporting groups
Arm/Group | Seroquel_XR | Chlorpromazine | Total
Number analyzed (Participants) | 194 | 190 | 384
Age Continuous [Mean (Standard Deviation); unit: years]
  age | 32.9 (10.70) | 32.0 (10.33) | 32.5 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 100 | 202
  Male | 92 | 90 | 182

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Positive and Negative Syndrome Scale (PANSS) Total Score at the End of Treatment at Day 42
Description: 6 weeks minus baseline.PANSS scale is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7. Total scores range 30-210 from better to worse.
Time Frame: Baseline and 6 weeks
Population: Per-protocol population was used as the analysis set for primary outcome, because this is a non-inferior design study.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 159 | 150
scores on a scale | -33.4 (1.45) [lower limit 1.45] | -35.9 (1.35) [lower limit 1.35]

2. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score at the End of Treatment at Day 42
Description: 6 weeks minus baseline PANSS scale is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7. 1 =Absent ,2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme The PANSS positive subscale score is the sum of the 7 positive item scores (ie, delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution and hostility) and ranges from 7 to 49. A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -9.9 (0.53) [lower limit 0.53] | -11.1 (0.51) [lower limit 0.51]

3. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score at the End of Treatment at Day 42
Description: 6 weeks minus baseline PANSS scale is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7. 1 =Absent ,2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme The PANSS negative subscale score is the sum of the 7 item scores (blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking), ranges from 7 to 49. A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -5.9 (0.5) [lower limit 0.50] | -6.7 (0.48) [lower limit 0.48]

4. Secondary Outcome: Change From Baseline in PANSS General Psychopathological Subscale Score at the End of Treatment at Day 42
Description: The PANSS psychopathological subscale score is the sum of 16 item scores(somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, active social avoidance), ranges from 16 to 112. A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -12.9 (0.74) [lower limit 0.74] | -13.9 (0.71) [lower limit 0.71]

5. Secondary Outcome: Change From Baseline in PANSS Aggression, Hostility Clusters Score at the End of Treatment at Day 42
Description: 6 weeks minus baseline PANSS scale is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7 (better to worse).
  1 =Absent ,2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -4.8 (0.33) [lower limit 0.33] | -5.4 (0.32) [lower limit 0.32]

6. Secondary Outcome: Change From Baseline in PANSS Depression Clusters Score at the End of Treatment at Day 42
Description: as for outcome 5
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -1.8 (0.18) [lower limit 0.18] | -1.7 (0.18) [lower limit 0.18]

7. Secondary Outcome: Number of Patients Achieving a Reduction of at Least 30% From Baseline PANSS Total Score at the End of Treatment at Day 42
Description: 6 weeks minus baseline PANSS scale is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7 (better to worse).Total scores range 30-210 from better to worse.
  1 =Absent,2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme.
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Number; unit: Percentage of participants
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
Percentage of participants | 57.7 | 66.3

8. Secondary Outcome: Percentage of Patients With Clinical Global Impression (CGI) Global Improvement Rating Less Than or Equal to 3 at the End of Treatment at Day 42
Description: 6 weeks minus baseline. The number of patients with CGI Global Improvement (CGI-I) rating at least "minimally improved" at the end of treatment at Day 42 was counted, and then got the proportion among all the patients.CGI-I is scored to rate the patient's change from baseline CGI on a seven-point scale (1="Very much improved", 7="Very much worse".)
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Number; unit: percentage of participants
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
percentage of participants | 87.6 | 88.9

9. Secondary Outcome: Change in the CGI Severity of Illness Score From Baseline at the End of Treatment at Day 42
Description: 6 weeks minus baseline The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale rating the severity of the patient's illness. The patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Baseline and 6 weeks
Population: Full analysis set was used for secondary outcome
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Number analyzed (Participants) | 194 | 190
scores on a scale | -1.8 (0.12) [lower limit 0.12] | -2.1 (0.11) [lower limit 0.11]

ADVERSE EVENTS:
Arm/Group | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) | Chlorpromazine
Serious Adverse Events (participants affected / at risk) | 0/196 | 2/192
Other Adverse Events (participants affected / at risk) | 142/196 | 166/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) (N=196) | Chlorpromazine (N=192)
Suicide Attempt (Psychiatric disorders) | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Fumarate (SEROQUEL) Extended-Release (XR) (N=196) | Chlorpromazine (N=192)
Constipation (Gastrointestinal disorders) | 49 | 31
Extrapyramidal Disorder (Nervous system disorders) | 17 | 58
Dizziness (Nervous system disorders) | 28 | 27
Insomnia (Psychiatric disorders) | 25 | 28
Agitation (Psychiatric disorders) | 24 | 21
Palpitations (Cardiac disorders) | 12 | 16
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Diarrhea (Gastrointestinal disorders) | 11 | 15
Tachycardia (Cardiac disorders) | 9 | 17
Heart rate increased (Cardiac disorders) | 8 | 15
Orthostatic Hypotension (Cardiac disorders) | 4 | 18
Hepatic Function Abnormal (Hepatobiliary disorders) | 11 | 9
Somnolence (Psychiatric disorders) | 15 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Akathisia (Nervous system disorders) | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other